CLINICAL TRIAL: NCT05145218
Title: A Multicenter, Randomized, Open, Parallel Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQB2450 Injection Combined With Androtinib Hydrochloride Capsules Versus Paclitaxel as Weekly Treatment in the Treatment of Recurrent Platinum-resistant Ovarian Cancer
Brief Title: A Clinical Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsules Versus Paclitaxel as Weekly Treatment of Relapsed Platinum-resistant Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-III-10
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Recurrent Platinum-resistant Ovarian Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 injection + Anlotinib Hydrochloride capsules (Experimental): TQB2450 injection: once every 21 days, 1200mg each time, intravenous infusion. The longest administration time should not exceed 24 months.
  Anlotinib Hydrochloride capsules: once a day, 12mg each time, oral administration on an empty stomach before breakfast for 2 weeks, withdrawal for 1 week, i.e. 3 weeks (21 days) as a course of treatment.
  Interventions: Drug: Anlotinib Hydrochloride Capsules; Drug: TQB2450 injection
- Paclitaxel injection (Active Comparator): 80mg/m2, intravenous drip, once a week (D1, D8, D15 of 21 days), 21 days as a course of treatment.
  Interventions: Drug: Paclitaxel injection

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsules — Anlotinib Hydrochloride is a multi-target tyrosine kinase inhibitor.
  Arms: TQB2450 injection + Anlotinib Hydrochloride capsules
Drug: Paclitaxel injection — Paclitaxel is a novel anti-microtubule agent.
  Arms: Paclitaxel injection
Drug: TQB2450 injection — TQB2450 is a programmed cell death protein 1 (PD-1) humanized monoclonal antibody.
  Arms: TQB2450 injection + Anlotinib Hydrochloride capsules

SUMMARY:
A clinical study to evaluate the efficacy and safety of TQB2450 injection combined with Anlotinib Hydrochloride capsules versus weekly treatment with paclitaxel of recurrent platinum-resistant ovarian cancer.A total of 405 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1) The subjects voluntarily joined the study, signed the informed consent form(ICF), and had good compliance;
* 2) age: 18-75 years old (when signing ICF; Eastern Cooperative Oncology Group (ECOG) Performance Status(PS) score 0-1; estimated survival time is more than 3 months;
* 3) Epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer confirmed by histopathology or cytopathology;
* 4) Subjects had disease recurrence or progression during prior chemotherapy with platinum-based regimens or within 6 months after the last dose of chemotherapy with platinum-based regimens (for at least 4 courses of treatment). Note: The definition of disease recurrence or progression needs to meet either of the following two items: a.Evidence of objective radiographic or clinical disease progression (for example, cytological reports of new ascites or pleural effusion); b.Persistent elevation of tumor marker CA125 (confirmed 1 week later) accompanied by clinical symptoms or physical examination indicating disease progression.
* 5) The number of previous chemotherapy regimens does not exceed 4 lines, and it is required that no more than 1 systemic treatment regimen is accepted after platinum resistance;
* 6) At least one measurable lesion was confirmed according toResponse Evaluation Criteria in Solid Tumors 1.1( RECIST 1.1) criteria;
* 7) The function of main organs are well and meet the following standards: (1) Routine Blood routine examination standards (without blood transfusion or correction with hematopoietic stimulating factor drugs within 7 days before the examination ): a) Hemoglobin（HGB） ≥90 g/L; b) Absolute value of neutrophil（NEUT）≥1.5×109/L; c) Platelets count（PLT）≥ 80×109/L. (2) The biochemical examination shall meet the following standards: a) Total bilirubin (TBIL) ≤ 2 times the upper limit of normal (ULN) (Patients with Gilbert syndrome ≤ 3 × ULN); b) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×ULN. If it is accompanied by liver metastasis, ALT and AST≤5×ULN; c) Serum creatinine (CR) ≤ 1.5×ULN or Creatinine clearance (CCR) ≥60ml/min (Cockcroft-Gault glomerular filtration formula). d）Serum albumin (ALB) ≥30g/L (no albumin supplement within 7 days). (3) Blood coagulation function or thyroid function test should meet the following standards:

  a) Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR)≤1.5×ULN (no anticoagulant therapy); b) Thyroid Stimulating Hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be examined. If T3 and T4 levels are normal, it can be selected. (4) Heart color Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.

  (5) Urine routine: urine protein <2+ (when the baseline urine protein ≥ 2+, the patient will undergo a 24-hour urine protein quantitative test within 7 days, and can only be selected when urine protein <1g);
* 8) Women must meet one of the following conditions:

  1. Surgical sterilization has been performed;
  2. For those who have been menopausal, the menopause has been stopped for at least 1 year; (3) Women with fertility must meet the following conditions: The serum pregnancy test before the first administration is negative and must be non-lactating subjects;During the entire study period, agree to use an approved method of contraception (for example: oral contraception, injection contraception or implanted, barrier contraception, spermicides and condoms, Intrauterine devices), and the method of contraception remained unchanged throughout the study period.

Exclusion Criteria:

* 1) Other malign combined diseases and medical history:

  1. Suffering from other non-epithelial ovarian tumors (for example, germ cell tumors, sex cord stromal tumors) or borderline ovarian epithelial tumors;
  2. Other malignant tumors appeared or were present within 3 years. The following two cases can be included: other malignant tumors treated by single operation have achieved 5-year DFS in a row; The cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  3. There are Multiple factors affecting oral medications (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.);
  4. Unrelieved toxic reactions higher than CTCAE level 1 caused by any previous treatment, excluding hair loss;
  5. Received major surgical treatment, open biopsy, or suffered obvious traumatic injury within 28 days before the start of the study treatment;
  6. Long-term unhealed wounds or fractures;
  7. Arterial/venous thrombosis events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage and cerebral infarction), deep vein thrombosis and pulmonary embolism, etc; (Prophylactic use of anticoagulant therapy is allowed for patients with thrombotic tendency or undergoing anticoagulant therapy.)
  8. Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders; i) Subjects with any severe and/or uncontrolled disease, including:

     1. After more than two kinds of drug treatment, blood pressure control is still not ideal (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg);
     2. Patients with grade ≥ 2 myocardial ischemia or myocardial infarction, arrhythmia (including corrected QT interval (QTc) ≥ 450ms (male) and QTc ≥ 470ms (female) and grade ≥ 2 congestive heart failure (New York Heart Association (NYHA) classification);
     3. Active or uncontrolled severe infection (≥ CTCAE grade 2 infection);
     4. Abnormal liver*:

        * Hepatitis B virus infection, HBsAg positive, HBV DNA positive or copy number exceeds the upper limit of normal value in the research center; Remarks: Continuous antiviral therapy (nucleoside analogues are recommended) and monitoring of HBV DNA every 3 to 6 months are recommended for HBsAg positive patients eligible for inclusion，HBcAb positive subjects but _HBsAg negative subjects can be monitored for HBV DNA every 3 to 6 months, and antiviral therapy is required if the virus is activated.
        * Hepatitis C virus infection, HCV antibody positive, HCV RNA positive or the test value exceeds the upper limit of the normal value of the research center; Remarks: Patients with HCV who are eligible for inclusion also need continuous antiviral therapy to prevent viral activation and can be monitored for HCV RNA every 3-6 months. If the virus is activated, direct antiviral therapy without interferon is recommended.
     5. Patients with renal failure requiring hemodialysis or peritoneal dialysis;
     6. Patients with a history of immunodeficiency, including Human Immunodeficiency Virus (HIV) positive or other acquired or congenital immunodeficiency disease, or with a history of organ transplantation;
     7. Previous or existing interstitial pneumonia, (non-infectious) pneumonia that requires adrenal corticosteroid therapy, currently suffering from other types of pneumonia ≥ 2, or lung function tests confirmed severely impaired lung function (Forced Expiratory Volume in the first second (FEV1) or diffusing capacity of lung for carbon monoxide ( DLCO) or DLCO per alveolar volume (DLCO /VA) accounts for the expected value %<40%) and other objective evidence;
     8. Poor control of diabetes (Fasting Blood Glucose (FBG) > 10mmol/L);
     9. Patients suffering from epilepsy and requiring medical treatment;
* 2) Tumor-related symptoms and treatment:

  1. Patients who had received surgery, chemotherapy, radiotherapy, hormone therapy, biotherapy, and immunotherapy within 4 weeks before the start of the study treatment (the washout period was calculated from the end of the last treatment); Patients who had previously received local radiotherapy could be included if they met the following conditions: The end of radiotherapy was more than 4 weeks after the start of study therapy (brain radiotherapy was more than 2 weeks); And the target lesions selected in this study are not in the radiotherapy area; Or the target lesion is located in the radiotherapy area, but progression is confirmed.
  2. Received the treatment of proprietary Chinese medicines with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions within 2 weeks before the start of the study treatment (Including compound cantharidin capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule, etc.);
  3. Previously received related immunotherapy drugs for programmed death-1 (PD-1), programmed death-Ligand 1 (PD-L1), cytolytic T lymphocyte-associated antigen-4 (CTLA-4) or similar Tyrosine Kinase Inhibitor (TKI) small molecule anti-angiogenesis drugs such as Androtinib Hydrochloride;
  4. Imaging (CT or MRI) shows that the tumor has invaded the periphery of important blood vessels or the investigator judges that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during the subsequent study;
  5. Patients with clinical symptoms of pleural effusion, pericardial effusion or ascites requiring Repeated puncture or drainage or those who have received drainage for the purpose of treatment within 1 month before randomization;
  6. Subjects with known Central Nervous System (CNS) metastasis and/or cancerous meningitis; Unless asymptomatic, or treated and stable, no radiographic evidence of new or enlarged brain metastases was found for at least 4 weeks after brain metastases treatment, and steroid or anticonvulsant therapy was discontinued for at least 14 days before study treatment began.
* 3) Study treatment related:

  1. Live attenuated vaccine vaccination history within 28 days before the start of the study treatment or planned live attenuated vaccination during the study period;
  2. Patients with a history of severe allergic disease and severe drug allergy.It is known to be allergic to any component prescribed in paclitaxel or TQB2450 injection or Anlotinib hydrochloride capsules prescription;
  3. Active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, corticosteroid or immunosuppressant) occurred within 2 years before the start of the study treatment. Replacement therapy (such as thyroxine, insulin, or physiological corticosteroid for adrenal or pituitary insufficiency, etc.) is not considered systemic therapy;
  4. Patients who have been diagnosed with immunodeficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (Dose>10mg/day prednisone or other curative hormones) and are still continuing to use them within 2 weeks of first administration; 4) Participated in other anti-tumor drug clinical trials within 4 weeks before grouping; 5) According to the investigator's judgment, subjects who have concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or who are considered unsuitable for inclusion in the group for other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival(PFS) evaluated by Independent Review Committee(IRC) | Baseline up to two years
  The period from the first use of the drug to disease progression or death (whichever occurs first);
Overall survival (OS) | Baseline up to two years
  The preriod from the first use of the drug to death from all causes. For subjects who are still alive at the last follow-up, the OS will be counted as data censored based on the last follow-up. For subjects who are lost follow-up, the OS will be counted as data cesored based on the last confirmed survival time before being lost to follow-up.

SECONDARY OUTCOMES:
Disease PFS evaluated by investigators | Baseline up to two years
  The period from the first use of the drug to disease progression or death (whichever occurs first)
PFS rate of 6 months: including PFS rate of 6 months evaluated by IRC and investigators; | Baseline up to six months
  The proportion of subjects reaching 6 months from firstly- recorded objective tumor response (complete remission(CR) or partial remission(PR)) to firstly-recorded objective tumor progression or death due to any cause (whichever occurred first) .
Objective response rate (ORR) evaluated by IRC and investigators | Baseline up to two years
  , the proportion of subjects whose tumors are evaluated as complete remission(CR) and partial remission(PR) by IRC and investigators. It is recorded from the first use of the drug to disease progression or initiation of a new anticancer treatment.
Duration of response (DOR) | Baseline up to two years
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first) .
Disease Control Rate (DCR) | Baseline up to two years
  Proportion of subjects whose tumors shrink or remain stable for a certain period, including complete remission（CR）, partial remission（PR） and stable disease（SD）;
OS rate of 12 months | Baseline up to one year
  The proportion of subjects who survive for 12 months after the first dose
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)，as well as abnormal laboratory examination indicators. | Baseline up to two years
  The proportion of AEs and SAEs recorded afte signing the informed consent form(ICF).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - AnYang Tumor Hospital, Anyang, Henan